CLINICAL TRIAL: NCT00951314
Title: Cocaine Dependence, Metabotropic Glutamate Receptor Subtype 5 (mGluR5) Density, Genetics and Craving
Brief Title: Brain Glutamate Receptors and Cocaine Dependence
Status: Terminated | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090188; 09-DA-0188
Record Dates: First submitted 2009-08-01; First posted 2009-08-04 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2013-03-19

CONDITIONS: Drug Abuse; Cocaine Dependence
Keywords: Genetic Polymorphisms; Metabotropic Glutamate Receptors; Positron Emission Tomograhy (PET); Cocaine Dependence; Cue-Induced Craving; Drug Abuse
MeSH Terms: conditions — Substance-Related Disorders; Cocaine-Related Disorders

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Objective:

Cocaine addiction continues to be an important public health problem with over 1.7 million users in the US alone. Cocaine addiction is characterized by compulsive drug use despite adverse consequences and high rates of relapse during periods of abstinence. Cocaine addiction may be mediated by neuroadaptations in reward-related learning and memory processes in the mesocorticolimbic dopamine system and glutamatergic corticolimbic circuitry. Metabotropic glutamate subtype 5 receptors (mGluR5) likely play essential roles in mediating some of the actions of drugs of abuse. Animal studies have shown that mGluR5 knock-out or blockade reduces self-administration of cocaine and cocaine-induced hyper-locomotion. However, to what extent mGluR5 are involved in the pathophysiology of cocaine addiction in humans is currently unknown, partly due to the lack of suitable methods to reliably quantify mGluR5 in the living human brain.

This protocol aims to determine whether the density of mGluR5 in brain is altered in participants with cocaine addiction compared to healthy controls using positron emission tomography (PET) and the recently developed radiotracer for mGluR5, [18F]SP203. We also aim to determine whether this density is related to genotype, history of cocaine use, and/or craving for cocaine.

Study Population:

The study populations will consist of healthy adults with no history of substance abuse and a matched group of healthy current primary cocaine dependent male and female participants (20-50 years old.; N=40/group).

Design:

Density of mGluR5 will be measured in cocaine dependent participants and healthy adults volunteers with PET and (18F)SP203, a radioligand with specificity for mGluR5. All participants will undergo genotyping to identify normal or variant mGluR5 gene associated with drug abuse. The intensity of craving for cocaine will be assessed while watching a video about cocaine use.

Outcome measures:

Density of mGluR5 will be compared between cocaine dependent participants and healthy controls. In addition, correlation among the genetic polymorphism, the craving response, and the density of mGluR5 will be determined.

DETAILED DESCRIPTION:
Objective:

Cocaine addiction continues to be an important public health problem with over 1.7 million users in the US alone. Cocaine addiction is characterized by compulsive drug use despite adverse consequences and high rates of relapse during periods of abstinence. Cocaine addiction may be mediated by neuroadaptations in reward-related learning and memory processes in the mesocorticolimbic dopamine system and glutamatergic corticolimbic circuitry. Metabotropic glutamate subtype 5 receptors (mGluR5) likely play essential roles in mediating some of the actions of drugs of abuse. Animal studies have shown that mGluR5 knock-out or blockade reduces self-administration of cocaine and cocaine-induced hyper-locomotion. However, to what extent mGluR5 are involved in the pathophysiology of cocaine addiction in humans is currently unknown, partly due to the lack of suitable methods to reliably quantify mGluR5 in the living human brain.

This protocol aims to determine whether the density of mGluR5 in brain is altered in participants with cocaine addiction compared to healthy controls using positron emission tomography (PET) and the recently developed radiotracer for mGluR5, [18F]SP203. We also aim to determine whether this density is related to genotype, history of cocaine use, and/or craving for cocaine.

Study Population:

The study populations will consist of healthy adults with no history of substance abuse and a matched group of healthy current primary cocaine dependent male and female participants (20-55 years old.; N=40/group).

Design:

Density of mGluR5 will be measured in cocaine dependent participants and healthy adults volunteers with PET and (18(F)SP203, a radioligand with specificity for mGluR5. All participants will undergo genotyping to identify normal or variant mGluR5 gene associated with drug abuse. The intensity of craving for cocaine will be assessed while watching a video about cocaine use.

Outcome measures:

Density of mGluR5 will be compared between cocaine dependent participants and healthy controls. In addition, correlation among the genetic polymorphism, the craving response, and the density of mGluR5 will be determined.

ELIGIBILITY:
* INCLUSION CRITERIA:

Cocaine dependent participants must meet DSM-IV criteria for cocaine dependence at the time of participation.

Control participants who provide appropriate matches for cocaine-dependent participants will be recruited on the following characteristics: age, and when possible, parental socio-economic status and/or years of parental education.

EXCLUSION CRITERIA:

Control Participants:

1. Psychiatric disease: DSM-IV criteria will be used (American Psychiatric Association, 1994). No subject with a current axis I diagnosis (except for nicotine dependence) will be allowed. Claustrophobia is also exclusionary.
2. History of Drug Abuse: Volunteers reporting current or having a significant history of illicit drug abuse will be excluded from the study. Subjects may use moderate amounts of alcohol and caffeine and smoke an occasional marijuana cigarette, but must not be dependent on alcohol, caffeine or marijuana. No alcohol or marijuana for at least 24 hours prior to scanning. No smoking after midnight on the night before a scan.
3. Current or Past Medication Use: Volunteers may not currently use chronic (daily for more than 10 to 14 days in the last month) prescription or over the counter medications, (including, but not limited to, anti-hypertensive, anti-allergy, pain). Over the counter or prescription medications may be used on an occasional basis (for treatment of self-limited conditions, such as occasional headache, musculoskeletal discomfort, allergic symptoms or pain). All medications will be discontinued at least 5 days before the experimental session.
4. CNS disease: History of known structural brain abnormalities (e.g., neoplasm, subarachnoid cysts), cerebrovascular disease, infectious disease (e.g., abscess), history of head trauma (defined as documented loss of consciousness > 5 min), history of seizures as an adult, sleep apnea, tic disorder.
5. Cardiovascular, pulmonary, or systemic disease: Repeated (measured on three separate occasions) diastolic blood pressure >90 mm Hg, or systolic blood pressure >135 mm Hg, known arrhythmia, symptomatic or known coronary artery disease; history of endocarditis, cerebral embolism, obstructive pulmonary disease, Factive tuberculosis, known endocrine disease (derangements in adrenal, thyroid, bone or reproductive function), known chronic renal or hepatic dysfunction, HIV seropositive, known current autoimmune disease involving the CNS.
6. Miscellaneous exclusionary criteria: Body weight greater than 300 lbs. Hematocrit < 39.0 for males or < 36.0 for females. Participants are also excluded if veins are inaccessible.
7. Radiation exposure: Any subject who has participated in any research studies in which he/she received a radiation exposure that would result in combination with the present study, in a total effective radiation exposure (from research studies) exceeding 5.0 rem in a year.
8. Novocain allergy or lack of bilateral ulner and radial arterial patency in subjects receiving arterial catheter as assessed by an Allen s test or Dopler test artery patency for all subjects to be catheterized.
9. Presence in body of metallic implants or materials that could be moved by the magnet of the MRI scanner: pacemakers, surgical implants, aneurism clips, dental braces, bullet(s) or other metallic materials. A history of working with metal with consequent possible metal fragments in the body.
10. Inability to lie flat for a few hours for the PET scans
11. Women who are pregnant or lactating and children under the age of 18 will be excluded to avoid unnecessary exposure to radiation to these populations.

Cocaine Dependent Subjects:

In addition to the exclusion criteria listed above with the exception of item i. b), subjects in this group will be excluded if:

1. They are actively seeking or engaged in substance abuse treatment. Justification: Videos viewed during this study may produce drug craving, producing a significant risk of relapse in a dependent individual attempting to remain abstinent. Any participant seeking treatment will be referred to treatment, since delaying entry into treatment to participate in a study unnecessarily increases exposure to the risks associated with active cocaine dependence. Assessment tool(s): Clinical interview at screening and repeat questioning at time of consent.
2. They are dependent on other substances except nicotine or cocaine at the time of participation. Use of other abused substances will be allowed as long as they are not currently dependent on any drug except nicotine and cocaine. Justification: Dependence on other substances may result in unique CNS deficits that would increase the noise in our data. Further, other dependence may contaminate neural processes examined. Nicotine dependence will be allowed since nicotine use is not associated with a drug high in normal usage and the prevalence of nicotine dependence in cocaine using individuals may make it impractical to exclude them. Assessment tool(s): Substance Use Disorders module of the SCID with confirmation by clinical interview and negative urine drug screen. Positive screens for cocaine are allowed.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07-14; Study Completion 2013-03-19

PRIMARY OUTCOMES:
Determine if cocaine dependent participants have a different mGluR5 density than healthy controls

SECONDARY OUTCOMES:
Determine if mGluR5 density in ventral striatum in cocaine dependent participants is associated with craving.

CONTACTS AND LOCATIONS:
Overall Officials: Alane Kimes, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States

REFERENCES:
- [Background] Ametamey SM, Kessler LJ, Honer M, Wyss MT, Buck A, Hintermann S, Auberson YP, Gasparini F, Schubiger PA. Radiosynthesis and preclinical evaluation of 11C-ABP688 as a probe for imaging the metabotropic glutamate receptor subtype 5. J Nucl Med. 2006 Apr;47(4):698-705. PMID 16595505
- [Background] Ametamey SM, Treyer V, Streffer J, Wyss MT, Schmidt M, Blagoev M, Hintermann S, Auberson Y, Gasparini F, Fischer UC, Buck A. Human PET studies of metabotropic glutamate receptor subtype 5 with 11C-ABP688. J Nucl Med. 2007 Feb;48(2):247-52. PMID 17268022
- [Background] Backstrom P, Hyytia P. Ionotropic and metabotropic glutamate receptor antagonism attenuates cue-induced cocaine seeking. Neuropsychopharmacology. 2006 Apr;31(4):778-86. doi: 10.1038/sj.npp.1300845. PMID 16123768